CLINICAL TRIAL: NCT02548728
Title: Oxytocin Treatment of Opioid Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-3041
Record Dates: First submitted 2015-07-21; First posted 2015-09-14 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-04

CONDITIONS: Opioid Dependence; Opioid Withdrawal
Keywords: Opioid Dependence; Opioid Withdrawal; Opioid; Oxytocin; OT (oxytocin); Intranasal administration
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): Self administration three times on the first day, then twice daily treatment with intranasal oxytocin spray for 4 days.
  Interventions: Drug: Intranasal Oxytocin Spray
- Placebo (Placebo Comparator): Self administration three times on the first day, then twice daily treatment with intranasal spray that does not contain oxytocin for 4 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin Spray — 10 insufflations (40IU of oxytocin total) given three times on day of enrollment and then twice daily for 4 days
  Other Names: Syntocinon spray
  Arms: Oxytocin
Drug: Placebo — 10 insufflations (40IU of placebo, same solution as active treatment minus oxytocin) given three times on day of enrollment and then twice daily for 4 day
  Arms: Placebo

SUMMARY:
Purpose: The purpose of this research study is to learn whether oxytocin treatment decreases use of and cravings for opioids (narcotics) in people who have been using opioids heavily for long periods of time and are unable to stop on their own.

Participants: Patients meeting DSM-IV-TR criteria for opioid dependence.

Procedures (methods): Subjects will have standard medications available for withdrawal symptoms from opioids and standard psychosocial interventions available in the inpatient setting. In addition, subjects will self-administer intranasal test treatments 3 times daily.

DETAILED DESCRIPTION:
The purpose of this research study is to learn whether oxytocin treatment decreases use of and cravings for opioids (narcotics) in people who have been using opioids heavily for long periods and are unable to stop on their own. Oxytocin is made naturally and is released in parts of the brain where it acts like a chemical signal from one cell to another. Oxytocin is approved by the Food and Drug Administration for stimulating labor in pregnant women but is not approved as a treatment for opioid dependence.

People who use large amounts of opioids every day or many days per week for weeks or months undergo chemical changes in their brains. They continue to use opioids frequently and heavily because, even though they may know opioid use is not good for their health, they have unpleasant experiences if they stop or decrease the amount used. Those experiences can include increased anxiety, difficulty sleeping, difficulty tolerating stress, and a craving to use opioids, as well as physical symptoms of withdrawal such as feeling sweaty or having chills, bone or joint aches, muscle cramps, nausea, diarrhea. Studies have shown that giving oxytocin to opioid-addicted animals diminished opioid use after they had been denied access to opioids for a while and reduced symptoms when they were put into opioid withdrawal.

This is a randomized, double-blind, Placebo-controlled trial in subjects with opioid dependence that will test the efficacy of intranasal Oxytocin (OT) treatment vs. Placebo (containing the same ingredients as the OT spray except OT) on:

1. reducing opioid withdrawal symptoms and
2. the total amount of standard, as needed (PRN) medications required to control withdrawal symptoms during medical opioid detoxification.

Treatment assignments will be random within each sex. Each treatment group will be composed of up to 25 subjects. Essentially, this study involves adding daily OT or Placebo administration on a fixed schedule onto standard symptom triggered treatment of opioid withdrawal using non-opioid medications.

Subjects will be recruited from patients admitted to the Addictions Detoxification Unit (ADU) at Wakebrook, the local mental health center for Wake County, NC for medical detoxification from opioids. There will be no selection on the basis of gender, ethnicity or race. ADU professional staff will be educated about inclusion and exclusion criteria for this study. They will describe the study to newly-admitted opioid-dependent patients who appear to meet criteria. If patients express interest in participation, ADU staff will either call the Study Coordinator (at UNC Hospitals) as soon as possible or inform a member of the research team who will visit the ADU each weekday morning. Also, research personnel will contact the ADU each morning and afternoon to inquire about newly admitted patients. If the Study Coordinator is contacted about a potential study candidate, the Coordinator will contact and inform the member of the research team who will visit ADU that morning about the potential study participant. As soon as possible after potential subjects are admitted to the ADU, research personnel will obtain informed consent and conduct an initial brief assessment to determine if subjects meet criteria for inclusion in the study.

The brief assessment includes completion of:

1. urine sample collection for rapid drug screen to confirm opioid use and to determine other current substance use and, in women, to test for pregnancy;
2. a review of medical exclusion criteria;
3. vital sign (VS) measurements;
4. the M.I.N.I. psychiatric interview screening questions for psychotic disorders, severe major depression, mania, and suicidality;
5. the Time Line Follow Back interview to quantify addictive substance consumption during the preceding 3 months;
6. the Structured Clinical Interview for DSM-IV (SCID) Substance Use Disorders Module to determine if prospective subjects meet DSM-IV-R criteria for opioid dependence, currently meet criteria for opioid withdrawal, and currently or in the past 3 months have met criteria for dependence on substances that are exclusionary for this study;
7. draw a 5-mL blood sample for serum sodium concentration assay. Physical examinations are completed by Wakebrook physicians within 24 hours after patients are admitted. Findings on physical examinations will not be available until later the day of admission or the following day, which will be after initiation of intranasal doses. If significant physical exam abnormalities are identified, treatments and further subject participation in the study will be stopped immediately. Vital signs are measured at regular intervals on these patients as part of clinical care. The investigators will draw blood to assay serum sodium concentrations as a safety measure for this study.

If need be, prospective subjects will receive PRN medications for withdrawal symptoms before recruitment procedures are initiated or intranasal test treatments are begun. Treatment Protocol and Measures: If subjects qualify for inclusion in the study, their withdrawal symptoms will be immediately measured using the well-validated Clinical Opiate Withdrawal Scale (COWS) and they will complete self-rating of opioid craving using a 100-mm visual analog scale (VAS), Subjective Opioid Withdrawal Scale (SOWS) and a baseline Spielberger State-Trait Anxiety Inventory (SSTAI). This will be followed by self-administration of their first intranasal dose of the substance to which they have been randomized under supervision of research personnel or ADU professional staff. The second dose on the first day of admission will be given 2 hours after the first. A third dose will be given later on the first day of admission (at least 4 hours after the second dose). On subsequent days of admission, doses will be taken twice daily (shortly before breakfast or lunch and dinner). All inpatient self-administration of intranasal test doses will be monitored by ADU or research staff. Each dose will consist of 10 insufflations of Syntocinon Spray or placebo (containing the same ingredients as Syntocinon Spray except for Oxytocin). Each insufflation given 30 sec apart and alternating between nostrils. Oxytocin and Placebo doses are administered from identical blind-labeled 60-ml spray bottles that deliver 0.1 ml of aerosolized solution/spray per insufflation. Intranasal test treatments will be administered for up to 5 days. After the first intranasal test dose, research personnel will complete the rest of the M.I.N.I. psychiatric interview. During the first 2 inpatient days objective COWS and subjective SOWS subject self-rating of opioid craving will be obtained every 4 hours or whenever subjects report or nurses observe the onset of withdrawal symptoms. Subsequently, the COWS and SOWS measures will be obtained twice daily or whenever withdrawal symptoms increase for at least 2 additional days and longer if subjects continue to exhibit significant symptoms. Subjects will complete the VAS subjective rating of opioid craving and the State portion of the SSTAI on each inpatient day starting on admission day 2 approximately 1 hour before their second intranasal test dose. In all subjects, per protocol, multiple as-needed non-opioid medications will be available for symptoms of opioid withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-45.
2. Regular opioid use (daily or nearly daily) for at least 6 months (subjective report).
3. Active DSM-IV diagnosis of opioid dependence.

Exclusion Criteria:

1. Meets DSM-IV criteria for dependence on psychoactive substances other than opioids, caffeine or nicotine within 6 months prior to screening.
2. Treatment with naltrexone in the last month.
3. History of a significant psychiatric illness including: lifetime history of mania requiring hospitalization, psychotic disorder, cognitive disorder; history during the last two years of eating disorder. Standing or as needed non-exclusionary medications for non-exclusionary psychiatric disorders will be permitted.
4. Unstable medical illness that could compromise consent to treatment, interfere with evaluation of study medication, or present a safety concern (e.g. uncontrolled diabetes mellitus, unstable hypertension, BMI <18 or >35, seizure disorder, traumatic brain injury, Parkinson's disease, AIDS). Adequately controlled conditions (such as diabetes mellitus, hypertension, asthma, HIV infection, and hepatitis C) will not be exclusionary. Standing or or as needed medications for non-exclusionary medical conditions will be permitted.
5. Serum sodium < 136 mEq/L (i.e., below the normal range) at the time of screening.
6. Significant abnormal findings on physical examination.
7. Women who are pregnant or breastfeeding.
8. In the judgment of the investigators, the individual would be considered a poor candidate.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cort A Pedersen, MD, Principal Investigator — University of North Carolina, Chapel Hill; James C Garbutt, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) in COWS Total Score on Days 1 to 5 Inclusive
Description: The Clinical Opiate Withdrawal Scale (COWS) is an 11-item, observer-rated tool for quantifying withdrawal symptoms. Each section is rated from 0 (no symptom) to 4 or 5 (most severe symptom). Total score is classified into a 4 point rating scale (mild 5-12, moderate 13-24, moderately severe 25-36 and severe more than 36 points). Lower scores are more favorable.
Time Frame: From days 1-5, the measure includes scores starting at time 0 through the maximal final time of up to 120 hours.
Measure: Mean (Standard Error); unit: Average COWS score * hours
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 6 | 6
Average COWS score * hours | 4.2 (1.5) | 3.4 (1.5)

2. Secondary Outcome: AUC in Subjective Opiate Withdrawal Scale (SOWS) Total Score on Days 1 to 5 Inclusive
Description: Least squares mean AUC day 1 pre-dose through Day 5 in SOWS; SOWS scores range from 0-64, with a lower score being more favorable
Time Frame: 5 days
Population: SOWS data not collected due to subject noncompliance in adhering to form completion.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: AUC in Visual Analog Scale (VAS) Score for Craving on Days 1 to 5 Inclusive
Description: Craving levels were measured using the VAS score on Days 1 to 5; the VAS scores range from 0 ("no cravings") to 100 ("most intense craving I have ever had"). Note that the value of AUC is a product of time multiplied by VAS scale score thus the numeric values are higher than the highest value on the scale.
Time Frame: Days 1-5, the AUC includes data starting from time 0 hours up to 120 hours post-dose.
Measure: Mean (Standard Deviation); unit: Average VAS score * hours
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 6 | 6
Average VAS score * hours | 1498 (839) | 2037 (2253)

4. Secondary Outcome: Speilberger State and Trait Anxiety Inventory
Description: The Spielberger State and Trait Anxiety Inventory (STAI) is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of state anxiety, which evaluates how the subject feels currently (transient anxiety). The State scale consists of 20 questions, each question rated 1-4, and a higher score indicates greater anxiety. Total score ranges from 20 (no anxiety) to 80 (maximum anxiety).
Time Frame: Daily up to 5 days
Population: STAI data not collected due to subject noncompliance in adhering to form completion.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxytocin (N=6) | Placebo (N=6)
Psychosis (Psychiatric disorders) | 1 | 0 — Two days after end of medication administration, subject developed paranoia and hallucinations while still in the detoxification unit, became agitated and was transferred to a hospital.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=6) | Placebo (N=6)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) — Difficulty falling asleep
Aching (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Chills (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal cramps (Gastrointestinal disorders) | 2 (2) | 2 (2)
Restlessnes (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4)
Sweats (General disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Restless legs (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes